CLINICAL TRIAL: NCT06008795
Title: Pterygopalatine Fossa (PPF) Block as an Opioid Sparing Treatment for Acute Headache in Spontaneous Subarachnoid Hemorrhage
Brief Title: BLOCK-SAH - PPF-Block for Post-SAH Headache
Acronym: BLOCK-SAH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); New York University (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB CED000000829; 1U01NS124613-01A1 (NIH)
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-05

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Headache
Keywords: Pterygopalatine Fossa Nerve Block
MeSH Terms: conditions — Subarachnoid Hemorrhage; Headache | interventions — Ropivacaine; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Sequential Parallel Comparison Design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 - Active - Active (Active Comparator): Subjects randomized to Group 1 will receive an active PPF nerve block in Stage 1 followed by an active PPF nerve block in Stage 2 of the Double-Blinded Trial Phase
  Interventions: Drug: Pterygopalatine Fossa Nerve Block with Ropivacaine and Dexamethasone
- Group 2 - Placebo - Active (Other): Subjects randomized to Group 2 will receive a placebo PPF-injection in Stage 1 followed by an active PPF nerve block in Stage 2 of the Double-Blinded Trial Phase
  Interventions: Drug: Pterygopalatine Fossa Nerve Block with Ropivacaine and Dexamethasone; Procedure: Placebo Pteryogpalatine Fossa Injection
- Group 3 - Placebo - Placebo (Placebo Comparator): Subjects randomized to Group 3 will receive a placebo PPF-injection in Stage 1 followed by a placebo PPF-injection in Stage 2 of the Double-Blinded Trial Phase
  Interventions: Procedure: Placebo Pteryogpalatine Fossa Injection

INTERVENTIONS:
Drug: Pterygopalatine Fossa Nerve Block with Ropivacaine and Dexamethasone — Each PPF-active nerve block will consist of 20mg (4ml) ropivacaine plus 4mg (1ml) dexamethasone
  Other Names: Pterygopalatine Fossa Nerve Block
  Arms: Group 1 - Active - Active; Group 2 - Placebo - Active
Procedure: Placebo Pteryogpalatine Fossa Injection — Each placebo PPF-injection will consist of 5ml normal saline
  Arms: Group 2 - Placebo - Active; Group 3 - Placebo - Placebo

SUMMARY:
BLOCK-SAH is a phase II, multicenter, randomized, double-blinded, placebo-controlled clinical trial with a sequential parallel comparison design (SPCD) of bilateral pterygopalatine fossa (PPF) injections with 20mg ropivacaine + 4mg dexamethasone (active, PPF-block) compared to saline (placebo) for headache in survivors of aneurysmal subarachnoid hemorrhage (SAH), while monitoring intracranial arterial mean flow velocities with transcranial Doppler (TCD) peri-intervention (intervention = PPF-injections: active or placebo)

ELIGIBILITY:
In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated ICF by participant or a legally authorized representative (LAR)
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged ≥18 and ≤ 85 years
4. Admitted with a primary diagnosis of spontaneous, non-traumatic, SAH within 72 hours of ictus hemorrhage
5. Disease-specific inclusion criteria:

   1. Spontaneous, non-traumatic SAH
   2. Subarachnoid pattern of hemorrhage warranting diagnostic DSA due to involvement of at least one of the following regions: quadrigeminal plate, prepontine cistern, perimesencephalic cistern, Sylvian fissure, or surrounding Circle of Willis
   3. Modified Fisher grade 1-4 (on presentation imaging)
   4. Hunt and Hess 1-3 or World Federation of Neurosurgeons grade 1-4 (on screening, included only if also fulfilling Glasgow Coma Scale verbal subscore ≥4)
   5. Minimum Glasgow Coma Scale verbal subscore of 4 (on screening)
6. Able to verbalize pain scale scores according to 11-point numeric pain scale

   In order to be enrolled and undergo randomization in this study, an individual must meet all of the additional criteria:
7. Stabilization period criteria:

   1. A minimum of 4 hours from DSA with clipping or coiling procedure (whenever applicable)
   2. Successful treatment of culprit vascular lesion (i.e., ≥90% obliteration of aneurysm), when applicable
8. Requiring a minimum of 15mg OME prn for headache analgesia during any 24-hour period during eligibility period

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Premorbid conditions:

   1. Pre-existing neurologic, psychiatric, or other condition that would confound neurologic assessment or would make difficult/impossible to accurately assess neurologic and/or functional outcome
   2. Pre-existing diffuse flow-limiting narrowing of arteries in the Circle of Willis, regardless of etiology (e.g., atherosclerosis, vasculitis, Moya-Moya syndrome)
   3. Prior use of opioid or barbiturate analgesics for at least two-thirds of the days in previous month, regardless of indication
   4. Diagnosis of substance use disorder in the previous year
   5. Infected or wounded skin, or a skin lesion at the site of puncture for PPF- injection
2. Uncorrected coagulopathy

   1. Platelet count < 50,000/μL, International Normalized Ratio (INR) > 1.7
   2. Requiring use of systemic anticoagulation and antiplatelet therapy (except for aspirin monotherapy).
3. SAH-specific:

   1. Head trauma as etiology of SAH
   2. Infection as cause for aneurysm or SAH (i.e., mycotic aneurysms)
   3. Inability to successfully treat culprit vascular lesion
   4. Diffuse vasospasm on pre-enrollment diagnostic CTA or DSA. Vasospasm is defined as moderate-to-severe arterial narrowing on DSA or CTA not attributable to atherosclerosis, catheter-induced spasm, or vessel hypoplasia, as determined by a neuroradiologist or neurointerventionalist
4. Standard pain regimen conditions

   1. Elevation of hepatic enzymes prohibiting use of scheduled APAP (i.e., AST or ALT > 3x upper limit level)
   2. Chronic liver condition with absolute contra-indication for APAP (even at lower maximum daily doses)
5. Participation in a concurrent investigational/interventional study (observational studies allowed)
6. Known to be pregnant, or with a positive pregnancy test
7. Allergy or intolerance to the medications used in the PPF-block (i.e., ropivacaine, dexamethasone) or standard pain regimen (APAP)
8. Vulnerable populations such as prisoners and inmates (abiding GCP per the study IRB)
9. Unable to receive first PPF-injection within 96 hours of ictus hemorrhage

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2023-12-17 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | within 24 hours after each PPF-injection spanning the 48 hours of double-blinded treatment period
  prn oral morphine equivalent (OME)/day use
Primary Safety Endpoint | at 48 hours from first PPF-injection (end of double-blinded treatment period)
  incidence of radiographic vasospasm
Primary Tolerability Endpoint | at 24 hours following the first PPF-injection
  rate of acceptance of second PPF-injection

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - University of Maryland Baltimore, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Albany Medical College, Albany, New York
  - University of Rochester Medical College, Rochester, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Oregon Health and Sciences University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Busl KM, Smith CR, Troxel AB, Fava M, Illenberger N, Pop R, Yang W, Frota LM, Gao H, Shan G, Hoh BL, Maciel CB; BLOCK-SAH Investigators. Rationale and Design for the BLOCK-SAH Study (Pterygopalatine Fossa Block as an Opioid-Sparing Treatment for Acute Headache in Aneurysmal Subarachnoid Hemorrhage): A Phase II, Multicenter, Randomized, Double-Blinded, Placebo-Controlled Clinical Trial with a Sequential Parallel Comparison Design. Neurocrit Care. 2025 Feb;42(1):290-300. doi: 10.1007/s12028-024-02078-z. Epub 2024 Aug 13. PMID 39138719